CLINICAL TRIAL: NCT01957891
Title: Effect of Induced Hypoxia at Multiple Wavelengths
Brief Title: Hypoxia at Multiple Wavelengths of Light
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP2552
Record Dates: First submitted 2013-09-19; First posted 2013-10-08 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Hypoxia in Healthy Individuals
Keywords: Hypoxia; Multiple wavelengths
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to assess the effect of progressive, incremental hypoxia at multiple wavelengths of light.

DETAILED DESCRIPTION:
No additional information is required.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 35 years of age
* Is American Society Anesthesiologist status 1
* Has a BMI between 18 and 30

Exclusion Criteria:

* Currently taking any medications other than birth control pills
* Has participate in an investigational drug study within one month prior to the start of the study
* Fails the Allen's Test to confirm patency of the colateral artery
* Subject is female with a positive pregnancy test, or is female and is unwilling to use effective birth control between the time of screening and study termination
* Has a positive urine continine or drug test
* Has an reported allergy to Lidocaine
* Has anemia or other hemoglobinopathy
* Has a room air saturation less than 95% by pulse oximetry
* Has an abnormal EKG
* Has an abnormal pulmonary function test via spirometry
* Is intolerant to a breathing mask apparatus
* Has a COHb greater than 3%, or MetHb greater than 2%
* Has another condition, which in the opinion of the principle investigator would not be suitable for participation in the study
* Is unwilling or unable to provide informed consent or comply with the study procedures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Assess the effect of progressive, incremental hypoxia at multiple wavelengths of light | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, MD, Principal Investigator — Duke University
Locations (1):
- HPPL Duke Univeristy, Durham, North Carolina, United States